CLINICAL TRIAL: NCT05681351
Title: An Open-Label Extension Study of Olezarsen (ISIS 678354) Administered Subcutaneously to Patients With Severe Hypertriglyceridemia (SHTG)
Brief Title: CORE-OLE: A Study of Olezarsen (ISIS 678354) Administered Subcutaneously to Participants With Severe Hypertriglyceridemia (SHTG)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 678354-CS15; 2022-501999-26-00 (Other: EU CTIS)
Expanded Access: NCT06360237 (Approved for marketing)
Record Dates: First submitted 2022-12-25; First posted 2023-01-12 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Severe Hypertriglyceridemia
Keywords: ISIS 678354; Olezarsen
MeSH Terms: conditions — Hypertriglyceridemia | interventions — olezarsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olezarsen (Experimental): Participants who completed either ISIS 678354-CS5 (NCT05079919) or ISIS 678354-CS6 (NCT05552326) study would be enrolled to receive olezarsen, subcutaneous (SC) injection, once every 4 weeks from Week 1 through Week 153.
  Interventions: Drug: Olezarsen

INTERVENTIONS:
Drug: Olezarsen — Administered as SC injection.
  Other Names: AKCEA-APOCIII-LRx; ISIS 678354

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of olezarsen in participants with SHTG.

DETAILED DESCRIPTION:
This is a multi-center, open-label extension (OLE) study of approximately 800 participants with SHTG who would be rolled over from studies ISIS 678354-CS5 (NCT05079919) or ISIS 678354-CS6 (NCT05552326). Day 1 of this study may be same as the Week 53 visit of either ISIS 678354-CS5 or ISIS 678354-CS6, as applicable. Participants will receive olezarsen during the 157-week treatment period. The study will include a 31-day qualification Period, a 157-week treatment period, and a 13-week post-treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

* Satisfactory completion of either ISIS 678354-CS5 or ISIS 678354-CS6 with an acceptable safety profile, per Investigator judgment. Satisfactory completion requires that the patient did not terminate early from treatment.
* Participants must be on a stable regimen of lipid-lowering therapy that should adhere to standard of care (SOC) per local guidelines. A patient may be eligible if their regimen of lipid-lowering therapy has been changed recently, provided that lipid lowering medications are optimized and stabilized for at least 4 weeks prior to the end of the Qualification Period of this OLE study; ideally, such changes are initiated after Week 53 of the index study (ISIS 678354-CS5 or CS6).
* A patient may re-enroll in the study after having completed the study when the Treatment Period was 53 weeks, if the patient satisfactorily completed the study with an acceptable safety profile, per Investigator judgment. In the case of re-enrollment, there is no limit on the time gap between completion of treatment under the previous protocol and dosing upon re-enrollment (i.e., may exceed 17 weeks between doses).

Key Exclusion Criteria:

• Have any new condition or worsening of existing condition which in the opinion of the Investigator would make the participant unsuitable for enrollment, or could interfere with the participant participating in or completing the study, including need for treatment with disallowed medications, or need to change the required stable regimen as per either ISIS 678354-CS5 or ISIS 678354-CS6 study entry criteria. It is acceptable to adjust a regimen of lipid-lowering therapy as described in the second Key Inclusion Criterion above, and it is acceptable to adjust or stop lipid-lowering therapy at or after Week 13 per Investigator judgment.

NOTE: Other Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 885 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants With Change in Clinical Laboratory Values From Baseline to Week 53, From Baseline to Week 105, and From Baseline to Week 157 | Baseline up to Week 157
Proportion of Participants Who Experience Adverse Events (AEs) | Baseline up to Week 157
Proportion of Participants Who Use Concomitant Medications | Baseline up to Week 157

CONTACTS AND LOCATIONS:
Locations (262):
- United States (65):
  - LA Universal Research Center, Inc., Los Angeles, California
  - University of California, San Diego (UCSD), San Diego, California
  - Metabolic Institute of America, Tarzana, California
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Finlay Medical Research, Greenacres City, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - Finlay Medical Research, Miami, Florida
  - Innovia Research Center, Inc., Miramar, Florida
  - Harmony Clinical Research, Inc., North Miami Beach, Florida
  - R & B Medical Center LLC, Tampa, Florida
  - VICIS Clinical Research, Tampa, Florida
  - JSV Clinical Research Study, Inc., Tampa, Florida
  - Bayside Clinical Research, Trinity, Florida
  - Centricity Research, Columbus, Georgia
  - IACT Health, Columbus, Georgia
  - Affinity Health, Oak Brook, Illinois
  - St. Vincent Medical Group, Inc., Carmel, Indiana
  - University of Kansas Medical Center (KUMC), Kansas City, Kansas
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - Louisville Metabolic and Atherosclerosis Research Center (L-MARC), Louisville, Kentucky
  - Grace Research, LLC, Bossier City, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - IRC Clinics, Towson, Maryland
  - Massachusetts General Hospital Heart Center, Boston, Massachusetts
  - University of Michigan- Endocrinology & Metabolism, Ann Arbor, Michigan
  - Aa Mrc, Llc, Flint, Michigan
  - Washington School of Medicine, St Louis, Missouri
  - Bryan Medical Center, Lincoln, Nebraska
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Hudson County Clinical Trials Research Center, Union City, New Jersey
  - Modern Medical, Brooklyn, New York
  - NYU Langone Health, Mineola, New York
  - Langone Medical Center, New York, New York
  - Vagelos College of Physicians and Surgeons of Columbia University, New York, New York
  - Orchard Park Family Practice, Orchard Park, New York
  - The Presbyterian Hospital DBA Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - Kenneth Hilty, Greensboro, North Carolina
  - Clinical Trials of America, LLC, Lenoir, North Carolina
  - Lexington, Winston-Salem, North Carolina
  - The Ohio State University, Columbus, Ohio
  - Central Oklahoma Early Detection Center, Edmond, Oklahoma
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Walker Family Care, Little River, South Carolina
  - Monument Health Clinical Research, Rapid City, South Dakota
  - Health Concepts, Rapid City, South Dakota
  - Chattanooga Research & Medicine, PLLC, Chattanooga, Tennessee
  - The Jackson Clinic, Jackson, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Juno Research, Houston, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Sante Clinical Research LLC, Kerrville, Texas
  - FMC Science, Lampasas, Texas
  - DCT- McAllen Primary Care, LLC, McAllen, Texas
  - Texas Institute of Cardiology, McKinney, Texas
  - SMS Clinical Research, LLC, Mesquite, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - Permian Research Foundation, Odessa, Texas
  - Diabetes & Glandular Disease Clinic, P.A., San Antonio, Texas
  - Tranquil Clinical and Research Consulting Services, Webster, Texas
  - Manassas Clinical Research, Manassas, Virginia
  - York Clinical Research, Norfolk, Virginia
  - WVU Heart and Vascular Institute, Morgantown, West Virginia
- Argentina (6):
  - CIPREC, Buenos Aires
  - Fundacion Favaloro, Buenos Aires
  - Centro Medico Dra. Laura Maffei-Investigacion Clinica Aplicad, Buenos Aires
  - Glenny Corp SA, Buenos Aires
  - Instituto Medico DAMIC, Córdoba
  - Clinica FUSAVIM Privada, Villa María
- Australia (5):
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Royal Adelaide Hospital, Adelaide
  - Royal Prince Alfred Hospital, Camperdown
  - Monash Medical Centre, Clayton
  - Dr Heart Pty Ltd, Woolloongabba
- Belgium (3):
  - Universite Libre de Brussels (ULB)- Hopital Erasme, Brussels
  - Jessa Ziekenhuis, Hasselt
  - Universitaire Ziekenhuizen Leuven, Leuven
- Brazil (7):
  - Centro Especializado em Cardiologia, Campinas
  - Nucleo de Pesquisa Clinica S/S, Curitiba
  - Hospital Universitario Walter Cantidio- UFC, Fortaleza
  - Nucleo de Pasquisa em Cirurgia Vascular, Porto Alegre
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo- FMUSP, São Paulo
  - Instituto do Coracao (InCor) do Hospital das Clinicas da FMUSP, São Paulo
  - CPQuali Pesquisa Clinica Ltda., São Paulo
- Bulgaria (26):
  - MHAT- Blagoevgrad AD, Blagoevgrad
  - Medical Center Doctor Staykov EOOD, Burgas
  - Medical Center Diamedical 2013 OOD, Dimitrovgrad
  - MHAT, Gabrovo
  - MHAT Haskovo AD, Haskovo
  - Multiprofile Hospital for Active Treament Pazardzhik, Cardiology Department, Pazardzhik
  - SBAL "Special Medic" Ltd., Plovdiv
  - UHMAT Kaspela Ltd, Plovdiv
  - University Multiprofile Hospital for Active Treatment Pulmed, Clinic of Endocrinology, Plovdiv
  - Medical Center Rusemed EOOD, Rousse
  - UMHAT Kanev AD, Rousse
  - DCC-1 Sliven Ltd., Sliven
  - Medical Center Smolyan Clinical Research OOD, Smolyan
  - Medical Center for Specialized Medical Help in Cardiovascular Diseases OOD, Sofia
  - UMHAT Tsaritsa Yoanna ISUL- Clinic of Cardiology, Sofia
  - Medical Center Endomedical, Sofia
  - Medical Center Kalimat EOOD, Sofia
  - MC Doctor Kalchev OOD, Sofia
  - Medical Centre Synexus Sofia, Sofia
  - UMHAT Sofiamed, Sofia
  - MHAT Silven to MMA Sofia, Sofia
  - Clinical of Cardiology, Stara Zagora
  - Medical Center Zara-Med, Stara Zagora
  - Diagnostic Consultative Center Equita (DCC Equita), Varna
  - Specialized Hospital for Active Treatment of Cardiology, Varna
  - Medical Centre "Nevromedics" EOOD, Veliko Tarnovo
- Canada (6):
  - Bluewater Clinical Research Group, Inc., Sarnia, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Clinique des Maladies Lipidiques de Quebec Inc., Québec, Quebec
  - Institut de Recherches Cliniques de Montreal, Montreal
  - Toronto General Hospital, Toronto
- Czechia (12):
  - MEDICUS SERVICES s.r.o., Brandýs nad Labem
  - University Hospital Hradec Králové, Hradec Králové
  - KardioBusak s.r.o., Louny
  - EDUMED s.r.o., Náchod
  - Fakultni nemocnice Ostrava, Ostrava
  - Vseobecna fakultni nemocnice, Prague
  - Fakultni Nemocnice v Motole, Prague
  - Praha Poliklinika Hurka, Prague
  - Endokrinologie Cerny Most s.r.o., Prague
  - Milan Kvapil s.r.o., Příbram
  - AeskuLab k.s, Teplice
  - MU Dr. Nina Zemkova s.r.o. Interni Ambulance, Uherské Hradiště
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Aarhus Universitet Hospital, Aarhus
  - Esbjerg Hospital, Esbjerg
  - Viborg Regional Hospital, Viborg
- Turku University Hospital, Turku, Finland
- France (9):
  - Louis Pradel Hospital, Bron
  - Chu Dijon Bourgogne, Dijon
  - Hôpitaux de Marseille, Marseille
  - Hopital Lapeyronie, Montpellier
  - AP-HP Hopital Pitie-Salpetriere, Paris
  - CHU de Nantes - Hôpital Nord Laennec, Saint-Herblain
  - CHRU de Strasbourg, Strasbourg
  - Groupement de Cooperation Sanitaire (GCS) ESLAN - Polyclinique Vauban, Valenciennes
  - GHM les Portes du Sud, Vénissieux
- Germany (4):
  - Charite- Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Forschungszentrum Ruhr, Witten
- Greece (2):
  - Evangelismos General Hospital Athens, Athens
  - Hygeia Hospital, Athens
- Hungary (8):
  - Lausmed Kft, Baja
  - DRC Gyógyszervizsgáló Központ Korlátolt felelősségű társaság Balatonfüred, Balatonfüred
  - Obudai Egeszsegugyyi Centrum, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Rakoczi Ferenc Korhaz, Miskolc
  - Dr. Vasas Szilard Haziorvosi Rendelo, Nyíregyháza
  - Kardiologia Szakrendeles, Nyíregyháza
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- India (2):
  - Vinaya Hospital and Research Centre, Mangalore
  - Sir Ganga Ram Hospital, New Delhi
- Israel (8):
  - Soroka Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (8):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXII, Bergamo
  - Policlinico di Sant'Orsola, Bologna
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specializzazione "Sant' Anna e San Sebastiano" di Caserta, Caserta
  - Ospdale E. Bassini, Milan
  - Asst Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera Universitaria Policlinico, Palmero
  - Department of Translational and Precision Medicine, Rome
- Lithuania (3):
  - Klinikiniai Sprendimai, UAB, Kaunas
  - Saules Seimos Medicinos Centras, Kaunas
  - Kardiologijos ir reabilitacijos klinika, UAB, Klaipėda
- Malaysia (2):
  - University Malaya Medical Centre (UMMC), Kuala Lumpur
  - Pulau Pinang Hospital, Pulau Pinang
- Mexico (3):
  - Scientia Investigacion Clinical Sc, Chihuahua City
  - Clinstile, S.A. de C.V., Mexico City
  - Centro de Investigacion Cardiometabolica S.C., Mexico City
- Netherlands (10):
  - Academic Medical Center, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Ziekenhuis Rijnstate, Arnhem
  - Het Van Weel-Bethesda Ziekenhuis, Dirksland
  - Ziekenhuis Gelderse Vallei, Ede
  - Bethesda Diabetes Research Center, Hoogeveen
  - Radboud UMC, Nijmegen
  - Erasmus MC, Rotterdam
  - University Medical Center Utrecht, Utrecht
  - Albert Schweitzer Ziekenhuis, Zwijndrecht
- New Zealand (2):
  - New Zealand Clinical Research, Auckland
  - Edgar Diabetes and Obesity Research Centre, Wellington
- The Lipid Clinic (Oslo University Hospital), Oslo, Norway
- Poland (11):
  - Uniwersytecki Centrum Kliniczne, I Klinika Kardiologii, Gdansk
  - Biokinetica Spolka Akcujna, Józefów
  - Centrum Medyczne Salvia, Katowice
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - Clinical Best Solutions, Lublin
  - ETG Lublin, Lublin
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan
  - Osrodek Badan Klinicznych Metabolica, Tarnów
  - Clinical Best Solutions Sp. z.o.o. Spolka Komandytowa, Warsaw
  - Przychodnia Futuremeds Wroclaw, Wroclaw
  - ETG Zamosc, Zamość
- Portugal (5):
  - Hospital Infante D. Pedro, Aveiro
  - Hospital COF Tejo, Lisbon
  - Hospital CUF Tejo, Lisbon
  - Centro Hospitalar Universitario De Sao Joao, Porto
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E., Santa Maria da Feira
- Cardioplus Center SRL, Baia Mare, Romania
- Slovakia (10):
  - Ambulancia diabetologicka a poruch latkovej premeny a vyzivy, Bratislava
  - Kardiologická ambulancia, Brezno
  - Cardio D&R, S.R.O. Kosice, Košice
  - Human-Care s.r.o., Košice
  - Vychodoslovensky Utsav srdcovych a cievnych chorob a.s., Košice
  - Interna a diabetologicka ambulancia- IN- DRA- s.r.o., Lučenec
  - Diab sro, Rožňava
  - Interna SK, s.r.o., Kardiologicka a interna ambulancia, Svidník
  - Nemocnica arm. generala L. Svobodu Svidnik, a.s, Svidník
  - Areteus sro, Trebišov
- South Africa (4):
  - Latros International, Bloemfontein
  - Medi Clinic Vergelegen, Cape Town
  - TREAD Research, Cape Town
  - University of Cape Town, Cape Town
- Spain (15):
  - Hospital Abente y Lago, A Coruña
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic De Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Jaen, Jaén
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Corporacio Sanitaria Parc Tauli- Hospital de Sabadell, Sabadell
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Virgen del Rocío, Seville
  - Hospital Universitari Sant Joan de Reus, Tarragona
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (2):
  - Sahlgrenska, University Hospital, Gothenburg
  - Karolinska University Hospital Huddinge, Stockholm
- Taiwan (5):
  - Kaohsiung Medical University Ching-Ho Memorial Hospital, Kaohsiung City
  - Mackay Memorial Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Shing Kong Wu Ho-Su Memorial Hospital, Taipei
- Turkey (Türkiye) (3):
  - Ege University School of Medicine, Department of Cardiology, Izmir
  - Necmettin Erbakan Universitesi Meram Tip Fakultesi, Konya
  - Hacettepe Üniversitesi Tıp Fakültesi, Sulhiye
- United Kingdom (9):
  - Centre for Diabetes, Endocrinology and Metabolic Disease, Woodhurst, Chatsworth
  - Huddersfield Royal Infirmary, Huddersfield, England
  - Waterloo Medical Care, Blackpool
  - Hull Royal Infirmiry, Hull
  - Oak Tree Surgery and Pensilva Health Centre, Liskeard
  - Manchester University NHS Foundation Trust, Manchester
  - Newquay Health Centre, Newquay
  - The Adam Practice, Poole
  - Sandwell and West Birmingham NHS Trust, West Bromwich

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/